CLINICAL TRIAL: NCT04365790
Title: Investigation of Gene Mutations or Changes in Protein Expression,as Biomarkers With Prognostic/Predictive Value, in Patients With Triple-negative and in Patients With HER2+ Breast Cancer Adenocarcinoma,Who Underwent Intensive Adjuvant Chemotherapy
Brief Title: Investigation of Gene Mutations in Patients With Triple-negative and Patients With HER2+ Breast Cancer Adenocarcinoma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hellenic Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: HE10/13
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
Keywords: Triple-negative breast cancer; HER2 positive breast adenocarcinoma
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with triple-negative breast cancer: Patients with histologically confirmed triple-negative breast cancer. Patients had been treated in Hellenic Cooperative Oncology Group (HeCOG)-affiliated departments of oncology
- Patients with HER2+ positive breast cancer: Patients with histologically confirmed HER2+ breast adenocarcinoma with high risk of recurrence. Patients had been treated in Hellenic Cooperative Oncology Group (HeCOG)-affiliated departments of oncology.

SUMMARY:
The present study is a transnational study in patients with high risk recurrent breast cancer who receive adjuvant chemotherapy with epirubicin and cyclophosphamide followed by docetaxel or paclitaxel.

DETAILED DESCRIPTION:
This will be a retrospective analysis of patients with histologically confirmed triple-negative or HER2+ operable breast cancer (with high risk of recurrence) who are treated at Hellenic Cooperative Oncology Group (HeCOG)- affiliated departments of oncology. Patients who participate are 18 years or older, women of any menopausal status with triple-negative or HER2+ breast cancer who receive epirubicin and cyclophosphamide every two weeks followed by docetaxel every three weeks or weekly paclitaxel. Patients with HER2-positive tumors are treated with trastuzumab, initiated concurrently with the first cycle of docetaxel, for 52 weeks. Pertuzumab may be combined with trastuzumab only in patients with node-positive disease.Patients can be treated with hormone therapy and/or radiotherapy. The investigation of the potential biomarkers will be performed using in situ methods in Formalin fixed paraffin embedded (FFPE) tumor sections. More specific will be investigated the expression of estrogen and progesterone receptors, the expression of SPARC proteins, special cellular activation and metastasis systems and other important pathways in cell life and reproduction.

Statistical analysis: The primary endpoint of the study will be the progression-free survival (PFS), defined as the time from treatment initiation to either the first documented disease progression or death from any cause. Second primary endpoint will be the overall survival (OS), defined as the time from treatment initiation to patient's death or last contact. Survival curves will be estimated using the Kaplan-Meier method and compared across groups with the log-rank test. The associations between the clinicopathological factors to be examined and the mortality rate will be evaluated with hazard ratios estimated with Cox proportional hazards model. The statistical analyses will be completed using the SAS software (SAS for Windows, version 9.3, SAS Institute Inc., Cary, NC).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Αny menopausal status is allowed
* triple-negative breast cancer
* HER2+ breast adenocarcinoma
* tumor size <= 5 cm
* presence of operable axillary lymph nodes or the presence of clinicopathological parameters indicating an intermediate or high risk of recurrence without the presence of infiltrated lymph nodes
* Performance status (PS) = 0 or 1
* adequate bone marrow function , heart, liver and kidney
* no other history of previous neoplasm or other serious illness

Exclusion Criteria: -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: This is a retrospective analysis of patients with histologically confirmed HER2- positive breast adenocarcinoma,triple-negative breast cancer with high risk of recurrence.
  Patients have been treated in Hellenic Cooperative Oncology Group (HeCOG)- affiliated departments of oncology.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2013-04-18 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From treatment initiation to the first documented disease progression, up to 5 years
Overall survival | from thee date of treatment initiation until death from any cause or date of last contact whichever occurred first, assessed up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: George Foutzilas, MD, Principal Investigator — Hellenic Cooperative Oncology Group
Locations (1):
- George Fountzilas, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Norton L. Theoretical concepts and the emerging role of taxanes in adjuvant therapy. Oncologist. 2001;6 Suppl 3:30-5. doi: 10.1634/theoncologist.6-suppl_3-30. PMID 11346683
- [Background] Fisher B, Bauer M, Wickerham DL, Redmond CK, Fisher ER, Cruz AB, Foster R, Gardner B, Lerner H, Margolese R, et al. Relation of number of positive axillary nodes to the prognosis of patients with primary breast cancer. An NSABP update. Cancer. 1983 Nov 1;52(9):1551-7. doi: 10.1002/1097-0142(19831101)52:93.0.co;2-3. PMID 6352003
- [Background] Nissen-Meyer R, Kjellgren K, Mansson B. Adjuvant chemotherapy in breast cancer. Recent Results Cancer Res. 1982;80:142-8. doi: 10.1007/978-3-642-81685-7_24. PMID 7036276
- [Background] Meyer JS, McDivitt RW, Stone KR, Prey MU, Bauer WC. Practical breast carcinoma cell kinetics: review and update. Breast Cancer Res Treat. 1984;4(2):79-88. doi: 10.1007/BF01806389. PMID 6378283
- [Background] Kononen J, Bubendorf L, Kallioniemi A, Barlund M, Schraml P, Leighton S, Torhorst J, Mihatsch MJ, Sauter G, Kallioniemi OP. Tissue microarrays for high-throughput molecular profiling of tumor specimens. Nat Med. 1998 Jul;4(7):844-7. doi: 10.1038/nm0798-844. PMID 9662379
- [Background] Skacel M, Skilton B, Pettay JD, Tubbs RR. Tissue microarrays: a powerful tool for high-throughput analysis of clinical specimens: a review of the method with validation data. Appl Immunohistochem Mol Morphol. 2002 Mar;10(1):1-6. doi: 10.1097/00129039-200203000-00001. PMID 11893029
- [Background] Camp RL, Charette LA, Rimm DL. Validation of tissue microarray technology in breast carcinoma. Lab Invest. 2000 Dec;80(12):1943-9. doi: 10.1038/labinvest.3780204. PMID 11140706